CLINICAL TRIAL: NCT04356391
Title: Efficacy of Pinhole Gum Rejuvenation Compared to Connective Tissue Graft in Treatment of Gingival Recession
Brief Title: Pinhole Surgical Technique Compared to Connective Tissue Graft in Treatment of Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Othman Shibly, Program Director of the Advanced Education Program in Periodontics, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00001141
Record Dates: First submitted 2020-01-29; First posted 2020-04-22 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Periodontal Diseases
Keywords: Gingival Recession; Marginal Gingiva; Root Coverage
MeSH Terms: conditions — Periodontal Diseases; Gingival Recession

STUDY DESIGN:
Intervention Model Description: Randomized, split-mouth, double blinded design clinical trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Connective Tissue Graft harvest from Palate (Active Comparator): In each participant, a tooth will be assigned to the Connective Tissue Graft (CTG) technique and another tooth to the Pinhole Technique. The tooth assigned to the CTG technique will receive the graft harvested from the palate.
  Interventions: Procedure: Connective Tissue Graft Technique
- collagen resorbable membrane material (Experimental): In each participant, a tooth will be assigned to the Connective Tissue Graft (CTG) technique and another tooth to the Pinhole Surgical Technique (PST). The tooth assigned to the PST technique will receive the collagen resorbable membrane material.
  Interventions: Procedure: Pinhole Surgical Technique

INTERVENTIONS:
Procedure: Connective Tissue Graft Technique — For the sites receiving the control technique (Connective Tissue Graft), the technique described by Langer B. and Langer L. will be started with a sulcular incision followed by a partial thickness flap. A CTG is then harvested according to the technique described by Bruno, the first incision is perpendicular to the 2nd premolar and 1st molar and is 2-3mm apical to their gingival margin as wide as the recipient site, followed by a second incision parallel to the for mentioned teeth, 1-2mm apical to the first incision, then the CTG is raised by periosteal elevator and released from apical and lateral attachments by sharp incision when needed. The graft is then prepared to have a homogenous thickness of 1.5-2mm. The donor CTG is stabilized to the underlying connective tissue interproximally using 4-0 Vicryl sutures. The recipient flap is repositioned coronally, to cover as much as possible of the graft with no tension, 2mm coronal to the CEJ, then sutured with 4-0 Vicryl sutures.
  Other Names: Graft Harvested from the Palate
  Arms: Connective Tissue Graft harvest from Palate
Procedure: Pinhole Surgical Technique — For the sites receiving the test technique (Chao Pinhole Surgical Technique) the surgery starts with a small pinhole opening in the alveolar mucosa apical to the mucogingival junction of the affected tooth, the flap is then undermined using special instruments to create a full thickness pouch, followed by extending the pouch horizontally and coronally to undermined the adjacent papilla without incising it and free the flap for its coronal displacement. Then multiple 2x12mm strips of collagen resorbable membrane material (Bio-Gide, Geistlich Pharma AG) are packed under the papilla to secure the flap in a coronal direction. Gentle pressure is applied for 5 minutes to minimize the thickness of the blood clot after each of the procedures. The patients are advised to brush all teeth and sites except the buccal surfaces of the operated-on teeth, which are to be cleaned with 0.12% Chlorhexidine mouth rinse.
  Other Names: Collagen Resorbable Membrane Material
  Arms: collagen resorbable membrane material

SUMMARY:
This study compares the efficacy of root coverage achieved by the Pinhole Surgical Technique (PST) technique and the Connective Tissue Graft (CTG) technique in the treatment of Miller class I and II gingival recession defects. All patients will receive PST in one quadrant and CTG in another quadrant.

The hypothesis being tested is: Pinhole Surgical Technique outcomes are not inferior to those of the Connective Tissue Graft surgical technique.

DETAILED DESCRIPTION:
Gingival recession is defined as the apical migration of the marginal gingiva and it leads to root surface exposure. It may be localized to a few sites or generalized to several teeth, and the severity may vary within the same person and between different people.

A variety of surgical techniques have been recommended to attain root coverage, including connective tissue graft, free gingival graft (FGG), pedicle flaps, double papilla grafts, coronally positioned flaps, coronal positioning of previously placed FGG, guided tissue regeneration (GTR), and the use of acellular dermal matrix (ADM), or enamel matrix derivatives. A recently developed technique used to attain root coverage is the Pinhole Surgical Technique (PST) described by Chao. This novel approach involves the separation of the gingiva and periosteum from the underlying bone with instruments inserted through a pinhole created in the vestibular area of the involved tooth while filling underneath the undermined interproximal papilla with strips of a bioresorbable membrane, rather than transferring gingival tissue from the palate to the area of recession. The advantage of this technique is the preservation of the gingival tissues and its blood supply, while freeing the flap from its apical attachment for ease of coronal displacement and adequate root coverage. In addition, the lack of a secondary surgical site may eliminate the accompanying pain and discomfort often reported in root coverage procedures.

The connective tissue graft technique was described by Langer and Langer in 1985, in which the patient's own connective tissue is taken mostly from the palate and used to cover the area of recession. The retro-molar pad area (tuberosity) has also been used because of the thickening of the sub-mucosa in that area. This graft material is carefully sutured into place and a coronally advanced flap placed and sutured over it, while part of the graft can be left exposed. Currently the connective tissue graft (CTG) is the most common and predictable treatment for gingival recession, and is considered the gold standard. Key advantages of the connective tissue graft procedure are the availability of two sources of blood supply to the graft: one from the recipient bed, and the other from the overlying flap, the perfect chromatic integration, an optimal esthetic outcome, and excellent color match. In addition, an increase in the thickness of the gingival tissues and the width of keratinized gingiva has been documented with the ability for creeping attachment which is not possible with the use of bioresorbable collagen membranes.

ELIGIBILITY:
Inclusion Criteria:

1. The patients should be above 18 years old.
2. The presence of Miller's class I or II gingival recession on at least two matching bilateral or contralateral gingival recession defects (≥ 2 mm).
3. Recession defect on maxillary incisors, maxillary and mandibular canines, or premolars.
4. Absence of a history of periodontal surgery at the involved sites in the last 12 months.
5. History of compliance with oral hygiene instructions and periodontal recall.
6. Sufficient palatal or tuberosity donor tissue thickness (> 2mm).

Exclusion Criteria:

1. Patients with systemic illness known to affect the outcome of periodontal therapy, including diabetes, immune deficiencies, etc.
2. Pregnant and lactating women
3. History of allergic reactions to drugs or materials used in the surgery including collagen.
4. Current use of any form of tobacco.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Change in (Complete root coverage determined by recession classification, percentage root coverage, and recession depth, Pain Index, Healing Index) is being assessed. | Postoperative: baseline, 6 weeks, 3, 6, 12, 18, and 24 months
  Complete root coverage (CRC): The number of sites that resulted in 100% root coverage.
Change in percentage root coverage is being assessed | Postoperative: baseline, 6 weeks, 3, 6, 12, 18, and 24 months
  Percentage root coverage (%RC): calculated as ([RD preoperative - RD postoperative]/RD preoperative) × 100%.
recession depth | 2 weeks preoperative
  Recession Depth (RD): Measured in millimeters from the gingival margin at the mid-buccal aspect of the root, to the Cemento-Enamel Junction (CEJ) or relative CEJ.
Change in Pain Index is being assessed | Postoperative: baseline, 6 weeks, 3, 6, 12, 18, and 24 months
  Pain index (PN): Pain is recorded on a horizontal pain scale of 0-10. Pain index as follows; Mild for ''0 to 3,'' moderate for ''4 to 6,'' and severe for ''7 to 10.''
Change in Healing Index is being assessed | Postoperative: baseline, 6 weeks, 3, 6, 12, 18, and 24 months
  Healing index (HI): A horizontal scale from 1-5 evaluating tissue color, response to palpation, granulation tissue, incision margin, suppuration, adopted from Aleksic. 1 (very poor). 2 (poor). 3 (good). 4 (very good).

SECONDARY OUTCOMES:
Change in periodontal parameters (clinical attachment level) is being assessed | baseline, 6 weeks, 3, 6, 12, 18, and 24 months postoperative
  Clinical attachment level (CAL): Measured in millimeters from CEJ or relative CEJ to the base of the periodontal sulcus at 6 sites per tooth.
change in periodontal parameters (probing depth) is being assessed | baseline, 6 weeks, 3, 6, 12, 18, and 24 months postoperative
  Probing depth (PD): Measured in millimeters from the gingival margin to the base of the periodontal sulcus at 6 sites per tooth.
change in periodontal parameters (width of keratinized tissue) is being assessed. | baseline, 6 weeks, 3, 6, 12, 18, and 24 months postoperative
  Width of the keratinized tissue (KTW): Measured in millimeters at mid-buccal aspect of the tooth from the gingival margin to the mucogingival junction.
Change in periodontal parameters (gingival thickness) is being assessed. | baseline, 6 weeks, 3, 6, 12, 18, and 24 months postoperative
  Gingival Thickness: Measured in millimeters at the mid-buccal of the gingiva and 2 mm apical the gingival margin at the attached gingiva or the alveolar mucosa using a #15 endodontic reamer with a silicon disk stop.
Change in periodontal parameters (gingival index) is being assessed. | baseline, 6 weeks, 3, 6, 12, 18, and 24 months postoperative
  Gingival index (GI): GI is measured according to Loe and Sillness and scored on a scale of 0 to 3.

CONTACTS AND LOCATIONS:
Overall Officials: Othman Shibly, DDS, Principal Investigator — University at Buffalo; Yahya Sayed Suliman Atassi, BDS, Study Director — University at Buffalo
Locations (1):
- 250 Squire Hall, Department of Periodontics, University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
If decided to share data, through publication in one of the journals, then it would include but not limited to statistical analysis, abstract, manuscript, consent forms, tables used for evaluations, and results.

REFERENCES:
- [Background] Miller PD Jr. A classification of marginal tissue recession. Int J Periodontics Restorative Dent. 1985;5(2):8-13. No abstract available. PMID 3858267
- [Background] Albandar JM, Kingman A. Gingival recession, gingival bleeding, and dental calculus in adults 30 years of age and older in the United States, 1988-1994. J Periodontol. 1999 Jan;70(1):30-43. doi: 10.1902/jop.1999.70.1.30. PMID 10052768
- [Background] Greenwell H, Fiorellini J, Giannobile W, Offenbacher S, Salkin L, Townsend C, Sheridan P, Genco R; Research, Science and Therapy Committee. Oral reconstructive and corrective considerations in periodontal therapy. J Periodontol. 2005 Sep;76(9):1588-600. doi: 10.1902/jop.2005.76.9.1588. PMID 16171452
- [Background] Langer L, Langer B. The subepithelial connective tissue graft for treatment of gingival recession. Dent Clin North Am. 1993 Apr;37(2):243-64. PMID 8477867
- [Background] Langer B, Langer L. Subepithelial connective tissue graft technique for root coverage. J Periodontol. 1985 Dec;56(12):715-20. doi: 10.1902/jop.1985.56.12.715. PMID 3866056
- [Background] Miller PD Jr. Root coverage using a free soft tissue autograft following citric acid application. Part 1: Technique. Int J Periodontics Restorative Dent. 1982;2(1):65-70. No abstract available. PMID 6959974
- [Background] Holbrook T, Ochsenbein C. Complete coverage of the denuded root surface with a one-stage gingival graft. Int J Periodontics Restorative Dent. 1983;3(3):8-27. No abstract available. PMID 6358084
- [Background] Grupe HE, Warren RF. Repair of Gingival Defects by a Sliding Flap Operation. Journal of periodontology 1956;27:92-95.
- [Background] Pfeifer JS, Heller R. Histologic evaluation of full and partial thickness lateral repositioned flaps: a pilot study. J Periodontol. 1971 Jun;42(6):331-3. doi: 10.1902/jop.1971.42.6.331. No abstract available. PMID 5282573
- [Background] Cohen DW, Ross SE. The double papillae repositioned flap in periodontal therapy. J Periodontol. 1968 Mar;39(2):65-70. doi: 10.1902/jop.1968.39.2.65. No abstract available. PMID 4870433
- [Background] Ross SE, Crosetti HW, Gargiulo A, Cohen DW. The double papillae repositioned flap--an alternative. I. Fourteen years in retrospect. Int J Periodontics Restorative Dent. 1986;6(6):46-59. No abstract available. PMID 3468092
- [Background] Bernimoulin JP, Luscher B, Muhlemann HR. Coronally repositioned periodontal flap. Clinical evaluation after one year. J Clin Periodontol. 1975 Feb;2(1):1-13. doi: 10.1111/j.1600-051x.1975.tb01721.x. PMID 1055724
- [Background] Allen EP, Miller PD Jr. Coronal positioning of existing gingiva: short term results in the treatment of shallow marginal tissue recession. J Periodontol. 1989 Jun;60(6):316-9. doi: 10.1902/jop.1989.60.6.316. PMID 2778599
- [Background] Sorrentino JM, Tarnow DP. The semilunar coronally repositioned flap combined with a frenectomy to obtain root coverage over the maxillary central incisors. J Periodontol. 2009 Jun;80(6):1013-7. doi: 10.1902/jop.2009.080553. PMID 19485834
- [Background] Tarnow DP. Semilunar coronally repositioned flap. J Clin Periodontol. 1986 Mar;13(3):182-5. doi: 10.1111/j.1600-051x.1986.tb01456.x. PMID 3457805
- [Background] Maynard JG Jr. Coronal positioning of a previously placed autogenous gingival graft. J Periodontol. 1977 Mar;48(3):151-5. doi: 10.1902/jop.1977.48.3.151. PMID 264963
- [Background] Al-Hamdan K, Eber R, Sarment D, Kowalski C, Wang HL. Guided tissue regeneration-based root coverage: meta-analysis. J Periodontol. 2003 Oct;74(10):1520-33. doi: 10.1902/jop.2003.74.10.1520. PMID 14653400
- [Background] Harris RJ. A comparative study of root coverage obtained with an acellular dermal matrix versus a connective tissue graft: results of 107 recession defects in 50 consecutively treated patients. Int J Periodontics Restorative Dent. 2000 Feb;20(1):51-9. PMID 11203548
- [Background] Chambrone L, Tatakis DN. Periodontal soft tissue root coverage procedures: a systematic review from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S8-51. doi: 10.1902/jop.2015.130674. PMID 25644302
- [Background] Chambrone L, Chambrone D, Pustiglioni FE, Chambrone LA, Lima LA. Can subepithelial connective tissue grafts be considered the gold standard procedure in the treatment of Miller Class I and II recession-type defects? J Dent. 2008 Sep;36(9):659-71. doi: 10.1016/j.jdent.2008.05.007. Epub 2008 Jun 26. PMID 18584934
- [Background] Henderson RD, Greenwell H, Drisko C, Regennitter FJ, Lamb JW, Mehlbauer MJ, Goldsmith LJ, Rebitski G. Predictable multiple site root coverage using an acellular dermal matrix allograft. J Periodontol. 2001 May;72(5):571-82. doi: 10.1902/jop.2001.72.5.571. PMID 11394391
- [Result] Chao JC. A novel approach to root coverage: the pinhole surgical technique. Int J Periodontics Restorative Dent. 2012 Oct;32(5):521-31. PMID 22754900

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT04356391/Prot_SAP_000.pdf